CLINICAL TRIAL: NCT04383366
Title: Agreement and Accuracy of Different Devices for the Measurement of Corneal Thickness and Corneal Curvature in Patients With Keratoconus
Brief Title: Agreement and Accuracy of Different Devices Corneal Measurements
Status: Completed | Type: Observational
Sponsor: Gerald Schmidinger (Other)
Responsible Party: Sponsor-Investigator, Gerald Schmidinger, Prof.Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: TOPOC
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with keratoconus
  Interventions: Device: Pentacam® (Oculus, Inc., Wetzlar, Germany); Device: Casia II (Tomey Germany, Nürnberg); Device: Spectralis Anterion (Heidelberg Engineering, Heidelberg, Germany)

INTERVENTIONS:
Device: Pentacam® (Oculus, Inc., Wetzlar, Germany) — Scheimpflug imaging
Device: Casia II (Tomey Germany, Nürnberg) — Anterior segment optical coherence tomography
Device: Spectralis Anterion (Heidelberg Engineering, Heidelberg, Germany) — Anterior segment optical coherence tomography

SUMMARY:
To compare repeatability, reproducibility and agreement of both, AS- OCT and Scheimpflug imaging, for the measurement of corneal curvature and corneal thickness in patients with keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 99 years
* Presence of keratoconus
* Signed informed consent

Exclusion Criteria:

* Contact lens history within 5 days
* Pathologic changes of the lid or conjunctiva on slit-lamp examination
* History of corneal ocular surgery/Previous corneal cross-linking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with keratoconus will be recruited in the outpatient department of the Department of Ophthalmology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
maximum K-value | 1 day

SECONDARY OUTCOMES:
Simulated minimum and maximum K-value | 1 day
Mean K-values | 1 day
Central Corneal thickness | 1 day
Thinnest corneal point | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Schmidinger, Prof.Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No